CLINICAL TRIAL: NCT00076206
Title: A Double-Blind, Parallel, Placebo-Controlled, Randomized Study to Evaluate the Efficacy and Safety of 3 Different Oral Dose Levels (1, 2, And 4 Mg) of CCI-779 in Subjects With Active Rheumatoid Arthritis on Concomitant Methotrexate Therapy
Brief Title: Study Evaluating CCI-779 in Active Rheumatoid Arthritis on Concomitant Methotrexate Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3066A3-206
Record Dates: First submitted 2004-01-15; First posted 2004-01-19 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — temsirolimus

ARMS (4):
- A (Experimental): CCI-779 1 mg dose to be taken orally daily up to 12 weeks.
  Interventions: Drug: CCI-779
- B (Experimental): CCI-779 2 mg dose to be taken orally daily up to 12 weeks.
  Interventions: Drug: CCI-779
- C (Experimental): CCI-779 4 mg dose to be taken orally daily up to 12 weeks.
  Interventions: Drug: CCI-779
- D (Placebo Comparator): Placebo dose to be taken orally daily up to 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CCI-779
  Arms: A; B; C
Drug: Placebo
  Arms: D

SUMMARY:
The primary objective of this study is to compare the therapeutic response and safety of 3 oral dose levels of CCI-779, with placebo in subjects with active rheumatoid arthritis (RA) who have been receiving stable doses of methotrexate (MTX) for at least 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Meet American College of Rheumatology (ACR) criteria for RA
* Have active RA consisting of ≥ 6 swollen and ≥ 6 painful joints
* ACR functional class I-III

Exclusion Criteria

* At screening the subject's prior medications are reviewed. (Prior history of disease-modifying antirheumatic drug (DMARD) use is recorded, including the start and stop dates of the most recently taken DMARDs)
* Significant concurrent medical diseases
* Abnormal chest radiograph, including findings consistent with interstitial pneumonitis, granulomatous disease, or pleural effusion and/or infiltration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer